CLINICAL TRIAL: NCT06257121
Title: A Pilot Study to Assess the Use of Surface-guided Radiotherapy in Head and Neck Cancer Patients Who Suffer From Anxiety
Brief Title: Comparing Radiotherapy Immobilization Systems for Anxious HNC Patients
Acronym: CRISP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Marie-Eve Pelland, Researcher, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-11940
Record Dates: First submitted 2023-12-19; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer; Claustrophobia; Anxiety
Keywords: Head and neck cancer; Anxiety; Claustrophobia; Surface-guided imagery; Radiation therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Claustrophobia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SGRT (Experimental): Patient position will be managed by optical surface management system (OSMS). Equipment for this procedure includes an IMRT board, a long head cushion (with transparent Timo, moldcare, and shim), anatomical markers the cushion (shoulders, under the chin, etc.), a kneefix and arm plates. Every day, prior to treatment, there will be (1) A lateral kilo voltage (kV) image for jaw positioning and (2) a CBCT with standard match (3D column then 3D GTV/PTV). During treatment, patients will undergo real-time monitoring with the VisionRT system (SGRT). A second CBCT will de carried mid-treatment (after the 2nd of 3 arcs) and patient's position will be adjusted if deemed necessary.
  Interventions: Device: OSMS position management

INTERVENTIONS:
Device: OSMS position management — Patient position management in real time during radiation using an optical Surface Management System (OSMS) (Vision RT)
  Other Names: VisionRT

SUMMARY:
Background: Radiotherapy is a mainstay of treatment for ENT cancers, and its indication is frequent. Patients are positioned and immobilized using a thermoplastic mask, which is attached to the treatment table for the duration of each daily treatment. The mask's purpose is to prevent patient movement and ensure reproducible positioning. The advantages of using thermoplastic masks come at a cost for many patients. It is well established that mask fixation and mask anxiety are major concerns for patients, adversely affecting their quality of life and hindering treatment compliance. Surface-guided radiotherapy (SGRT) enables patients to be positioned and their movements monitored in real time during treatment. This technique has become more widely available in recent years, and is attractive because it does not involve ionizing radiation. However, although preliminary data have suggested a potential reduction in anxiety, this technique has not been evaluated for ENT RT in anxious/claustrophobic patients who cannot tolerate immobilization masks.

Objective: Investigators propose a pilot study to evaluate the feasibility and tolerability of using SGRT to manage position for patients with ENT cancer who report claustrophobia/anxiety.

Methodology: 15 participants will be recruited by the treating radiation oncologist from among patients scheduled to undergo radiation therapy at CHUM for their ENT cancer and identifying as claustrophobic/anxious. Participants who consent will be scheduled to undergo their radiotherapy using SGRT. Patients will be systematically treated with Volumetric Modulated Arc Therapy (VMAT) using SGRT on the linear accelerator with the Optical Surface Management System (OSMS) for the duration of the radiotherapy.

Measures: Patients' anxiety will be assessed using the GAD-7 and the CLQ throughout the treatment process. The feasibility and accuracy of radiotherapy treatment will be assessed using planning and daily pre-treatment examinations. In addition, skin toxicity will be assessed weekly.

Analyses: 1) Descriptive analyses, i.e. frequencies for categorical variables and means and standard deviations for continuous variables. 2) Estimation of confidence intervals.

Anticipated outcomes: Completion of this pilot project will enable investigators to plan and refine the methodological and organizational aspects for a large-scale study, i.e., a Phase III clinical trial comparing the use of SGRT with the use of a thermoplastic immobilization mask for anxious patients.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older
* Able to fluently speak, read and write French or English
* Histologically confirmed head and neck cancer
* Patients treated with radiotherapy as primary treatment
* Identified as having moderate mask anxiety / claustrophobia (i.e. a score of 10 or more on the Generalized Anxiety Disorder 7 item (GAD-7) questionnaire and / or a score of 28 or more on the Claustrophobia questionnaire (CLQ) suffocation subscale and / a score of 24 or more on the CLQ restriction subscale
* An Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0-2
* Able to understand and sign consent form
* Patients must be willing to comply with treatment plan and other study procedures

Exclusion Criteria:

* Patients with significantly altered mental status or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study
* Patients who cannot stay still during fraction because of a disorder (e.g., Parkinson's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety questionnaire | weekly from baseline to last week of treatment
  Generalized Anxiety Disorder Questionnaire (GAD-7), GAD-7 total score for the seven items ranges from 0 to 21. Higher score indicates worse outcome.
Anxiety behavior | weekly from baseline to end of radiation therapy, an average of 7 weeks
  Behavioral assessments of anxiety: (a) use of psychoactive (anxiolytic) medication; (b) use of psychological interventions / strategies (exposure therapy, relaxation / meditation, etc.); (c) use of music in treatment room; (d) need for vocal reassurance by technologists during scan/MRI; (e) exam interruptions
Claustrophobia | weekly from baseline to end of radiation therapy, an average of 7 weeks
  Claustrophobia Questionnaire (CLQ), includes two subscales of 14 and 12 items, total scores range from 0 to 104. Higher score indicates worse outcome.

SECONDARY OUTCOMES:
Well-being | weekly from baseline to end of radiation therapy, an average of 7 weeks
  Functional Assessment of Cancer Therapy scale (FACT-G7). Total score for seven items ranges from 0 to 28. Higher score indicates better outcome.
Setup consistency | Once - at treatment planning, on average 2 weeks after baseline
  Setup consistency between consecutive treatment planning scans
Intrafraction setup consistency | Daily from first to last radiotherapy treatment fraction, an average 7 weeks.
  Intrafraction setup consistency as reported by the surface guidance system (total amplitude & max deviation over time)
Fraction time | Daily from first to last radiotherapy treatment fraction, an average 7 weeks.
  Daily total fraction time as recorded
Skin toxicity | weekly from baseline to end of radiation therapy, an average of 7 weeks
  Skin toxicity grade assessed by treating rdio-oncologist at weekly follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve Pelland, Ph.D., Principal Investigator — CHUM

IPD SHARING:
Plan to Share IPD: No